CLINICAL TRIAL: NCT06880068
Title: Validity and Reliability of the Dual Task Impact on Daily Living Questionnaire in Patients with Parkinson's Disease
Brief Title: Reliability and Validity of DIDA-Q in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MarmaraU-SANLI-ERSOZ-001
Record Dates: First submitted 2025-01-13; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Dual-task Assessment; Neurological Physiotherapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Dual Task Impact on Daily-living Activities Questionnaire — This questionnaire makes us assess dual-task performance while performing daily-living activities.

SUMMARY:
The aim of our study is to investigate the validity and reliability of the Dual Task Impact on Daily-living Activities (DIDA-Q) to assess the degree of difficulty felt when performing dual tasks during activities of daily living in patients with Parkinson's disease. In our study, the validity and reliability of a questionnaire to assess the degree of difficulty felt while performing dual tasks during activities of daily living in Parkinson's Disease will be examined for the first time. The study will include 95 participants with Hoehn-Yahr Stage 1-3, diagnosed with Idiopathic Parkinson's Disease and able to walk 10 metres without an assistive device.

DETAILED DESCRIPTION:
Dual task ability is defined as the ability to perform two activities simultaneously . It is known that the ability to perform a motor or cognitive secondary activity at the same time during walking (talking to a person next to you while walking or carrying objects while walking) leads to gait and balance problems of different severity depending on the type of secondary task in Parkinson's Disease (PD). When patients with Parkinson's Disease (pwPD) are exposed to dual-task walking, their walking speed and length of stride decrease, and the frequency of freezing phenomena during walking increases. Consequently the risk of falling increase during activities of daily living. Individuals often perform dual tasks while performing activities of daily living because of the nature of the tasks' requirements. Therefore, it has become important to evaluate dual task performance in order to create the right treatment plan in the field of neurological physiotherapy and rehabilitation. Although dual task performance is evaluated with different formulae in the literature, the number of scales evaluating the level of difficulty perceived by the patient during the performance of activities of daily living under dual task is limited. The validity of the existing scales for PD has not been studied. The Dual-task Impact on Daily-living Activities Questionnaire (DIDA-Q) is a patient-reported questionnaire developed to assess the degree of difficulty perceived when performing dual tasks during activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Idiopathic Parkinson's Disease according to UK Brain Bank criteria
* Walking at least 10 metres without an assistive device
* To have the cognitive capability to understand and answer the questions asked in the scale

Exclusion Criteria:

* Having any neurological disease other than idiopathic Parkinson's Disease
* The person has an orthopaedic or cardiopulmonary disease that affects walking
* Severe hearing-visual impairment

Ages: 39 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed with Parkinson's disease were included.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2024-01-13 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
DIDA-Q | 1 week
  Dual Task Impact on Daily-living Activities Questionnaire, higher scores means bad dual task performance

OTHER OUTCOMES:
Six Spot Step Test cognitive | 1 week
  Designed to assess motor-cognitive dual task performance.
Dual Task Interference | 1 week
  It is calculating with a formula which contain single and dual task performance.
Dual Task Questionnaire | 1 week
  patient-reported questionnaire used to measure dual-task performance
Parkinson Activity Scale | 1 week
  a scale to assess patients' mobility and transfers
Mini-Mental State Examination | 1 week
  a short questionnaire giving information about the cognitive status of the patients
Freezing of Gait Questionnaire | 1 week
  a scale questioning the frequency of freezing and freezing qualities in walking

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Faculty of Medicine, Istanbul, Çapa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No